CLINICAL TRIAL: NCT06006039
Title: An Explorative Study to Examine the Role of IL-23-Responsive Immune Cell Subsets in Post-Operative Recurrence in Patients With Crohn's Disease.
Brief Title: The Role of IL-23-Responsive Immune Cell Subsets in Post-Operative Recurrence in Patients With Crohn's Disease.
Acronym: DIVE-23
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Geert D'Haens, prof dr G.R.A.M. D'Haens, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL82888.018.22
Record Dates: First submitted 2023-07-12; First posted 2023-08-23 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Crohn´s Disease
Keywords: Crohn's Disease; Interleukin-23; Postoperative recurrence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The investigators will retain mucosal biopsies and blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory Bowel Diseases (IBDs), including ulcerative colitis and Crohn's disease (CD), constitute a group of debilitating chronic diseases that profoundly impact patient quality of life and incurs large costs in terms of treatment and lost productivity. Incidence of IBD is rising worldwide, and there is a pressing clinical need for development of new therapies. Discovery and development of effective therapies to treat IBDs depend first on a better understanding of the underlying mechanisms, including how proinflammatory cells proliferate unchecked.

It has been established that the cytokine interleukin (IL)-23 plays a pivotal role in IBD pathophysiology and antibodies targeting IL-23 are currently in late stage development for the treatment of both CD and ulcerative colitis (UC). IL-23 is part of the IL-12 family of cytokines (which includes IL-12, IL-27 and IL-35). The p40 subunit is shared among IL-23 and IL-12; the p19 subunit is unique to IL-23. Thus far, the efficacy of selective anti-IL-23 blockade (via anti-p19 antibodies) appears 5-10% better with respect to clinical and endoscopic outcomes than targeting both IL-23 and IL-12 using anti-p40 antibodies. Understanding the effects of IL-23 (and IL-12) in IBDs requires identification of the most relevant immune cells that respond to these cytokines. One likely cell type controlled by the IL-23 pathway are innate lymphoid cells (ILCs). ILC3s (a subset of ILCs) are dominant in healthy intestinal tissue and capable of producing IL-22 which maintain intestinal epithelial homeostasis. Disturbances in the amounts of IL-22 caused by changes in the stimulatory cytokine IL-23 in tissues, may therefore cause inflammatory responses. IL-23 may facilitate the IL-12-induced shift of ILC3s to ILC1s which are contributing to the disease-causing chronic inflammation.

The DIVE 23 project is designed to understand the role of IL-23 in human IBD, in particular CD. It is hypothesized that IL-23R+ cells in the gut, are drivers of chronic inflammation in CD and determine the impact of IL-23 inhibition. To this end the investigators plan to extensively characterize the IL-23-responsive cell populations in inflamed and non-inflamed intestinal tissues of CD patients with postoperative recurrence in order to identify IL-23-responsive immune cell populations that are associated with disease activity. Patients will be treated in routine medical practice with biological agents and will undergo a second ileocolonoscopy 12-16 weeks later to investigate the impact of the different interventions on the mucosal immunology driving CD.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years;
* Male or non-pregnant, non-lactating females;
* Patients with postoperative recurrence at routine endoscopy 6-24 months following resection, defined by presence of ulcerations (endoscopic Rutgeerts' score >i2a) in the neoterminal ileum;
* In the opinion of the investigator, the subject is capable of understanding and complying with protocol requirements;
* The subject signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

* Any conditions (eg, history of alcohol or substance abuse, or lack of compliance) which, in the opinion of the investigator, may interfere with the patient's ability to comply with study procedures;
* Any condition in which one of the potential treatments are contraindicated in the opinion of the investigator (eg, cardiac failure class 3-4 according to the New York Heart Association [NYHA], multiple sclerosis, active infections).
* Received any investigational drug in the past 30 days or 5 half-lives, whichever is longer.
* Currently participating or planning to participate in a study involving an investigational product.
* Active or planned pregnancy during the study.
* Prior diagnosis of dysplasia in the colon (excluding in resected adenomas).
* History of malignancy in the 3 years prior to randomization except for non-melanoma skin cancer.
* Received a biologic treatment between surgery and first endoscopy.
* Positive Clostridium difficile toxin B in faeces. Patients who test positive can be treated per local practice and still enter the study if no longer than 4 weeks after the screening visit, they test negative for Clostridium difficile toxin B.
* Presence of a stoma without ileocolonic anastomosis or pouch.
* Active perianal abscess or draining fistula
* ALT or AST > 3x the upper limit of normal measured at screening
* Increased risk of bleeding: coagulation disorder, use of anticoagulants and DOACs

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be performed in CD patients with postoperative recurrence. Patients will be counselled prior to their routine endoscopy (typically 6-9 months after surgery). In practice, this will be approximately be between one and two weeks before the routine endoscopy. The investigators intend to evaluate 20-30 patients for this study and recruit 40 patients. The reason for this, is that there is a possibility that patients do not have enough inflammation (Rutgeerts ≤i2a) and therefore cannot be included.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes in concentration and amounts of IL-23 responsive cells in postoperative CD at baseline endoscopy and after 12-16 weeks of routine care treatment with a biological agent. | Week 16
  Single cell analysis

SECONDARY OUTCOMES:
Changes in concentration and amounts in IL-23 pathway cytokines and mediators, at baseline and after 12-16 weeks of biological treatment. | Week 16
  Single cell analysis
Change in modified Rutgeerts' score at baseline endoscopy and follow-up endoscopy (12-16 weeks after biological treatment) | Week 16
  Endoscopic outcome measurement
Change in SES-CD score at baseline endoscopy and follow-up endoscopy (week 12-16, after biological treatment) | Week 16
  Endoscopic outcome measurement
Change in the Harvey-Bradshaw Index (HBI) score at baseline visit and follow-up visits at week 8 and week 12-16. | Week 16
  Clinical outcome measurement
Change in Robarts histopathology index (RHI) score at baseline endoscopy and follow-up endoscopy (week 12-16, after biological treatment). | Week 16
  Histology outcome measurement

CONTACTS AND LOCATIONS:
Locations (2):
- Mount Sinai, Toronto, Ontario, Canada
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided